CLINICAL TRIAL: NCT05445960
Title: Correlation Between Intraoperative Tourniquet Use and Limb pH, Functional Measures and Patient-reported Outcomes After Ankle Fracture Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Lara Atwater, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00022560
Record Dates: First submitted 2022-05-10; First posted 2022-07-06 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Ankle Fractures; Ankle Fracture - Lateral Malleolus; Ankle Fracture, Bimalleolar; Ankle Fracture, Trimalleolar; Ankle Fracture - Medial Malleolus; Maisonneuve's Fracture; Syndesmotic Injuries; Fibula Fracture
MeSH Terms: conditions — Ankle Fractures; Fibula Fractures; Ankle Injuries | interventions — Tourniquets

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tourniquet (Active Comparator): This arm will have a tourniquet placed around the thigh inflated to 250mmHg for the duration of surgery (until splint placed) or 2 hours, whichever is shorter, during ankle fracture surgery.
  Interventions: Procedure: Tourniquet
- No Tourniquet (No Intervention): This arm will have a tourniquet placed around the thigh but NOT inflated for the duration of ankle fracture surgery.

INTERVENTIONS:
Procedure: Tourniquet — This arm will have a tourniquet placed about the thigh and inflated to 250mmHg for the duration of ankle fracture surgery or 2 hours, whichever is shorter.
  Arms: Tourniquet

SUMMARY:
This study aims to 1) characterize skeletal muscle pH during/after tourniquet use and 2) investigate any relationship between intraoperative tourniquet use and postoperative functional measures and patient-reported outcomes.

DETAILED DESCRIPTION:
Tourniquets are widely accepted as "safe" for up to two hours of continued use, despite known risks and a paucity of literature supporting this duration. Complications of tourniquets include tourniquet site pain, increased surgical site pain and swelling from reperfusion, neuropraxia, vascular injury, functional weakness, and decreased muscle endurance. Similar to compartment syndrome, tourniquets eliminate the tissue perfusion gradient necessary for oxygen, glucose, and lactic acid exchange. Lack of molecular exchange within the tissue is thought to result in tissue anoxia and acidosis, leading to cellular death of skeletal muscle and nerves. This study randomizes patients undergoing ankle fracture surgery to tourniquet or no-tourniquet arms and studies outcomes including continuous intramuscular pH during and after surgery, and patient-reported outcomes and functional measures up to 3 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years to 89 years) undergoing surgical ankle fracture fixation at OHSU

Exclusion Criteria:

* sepsis
* other significant long bone or internal injuries (including ipsilateral limb injuries).

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2021-08-17 (Actual); Primary Completion 2026-03-17 (Estimated); Study Completion 2027-03-17 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Patient-Reported Outcomes Measurement Information System Physical Function Subscale at 12 Weeks | Collected preoperatively and 12 weeks postoperatively
  Patient-Reported Outcomes Measurement Information System (PROMIS) Physical Function (PF) subscale, a Patient Reported Outcome survey used widely in orthopaedic literature, will be obtained and reported in points. For PROMIS measures, higher scores equals more of the concept being measured (e.g., more Fatigue, more Physical Function). A score of 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For example a score of 40 is one SD lower than the mean of the reference population where as a score of 60 is one SD higher than the mean of the reference population. Thus a score of 60 is one standard deviation above the average referenced population. This could be a desirable or undesirable outcome, depending upon the concept being measured.
Change from Baseline Patient-Reported Outcomes Measurement Information System Pain Interference Subscale at 12 weeks | Collected preoperatively and 12 weeks postoperatively
  Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference (PI) subscale, a Patient Reported Outcome survey used widely in orthopaedic literature, will be obtained and reported in points. A score of 50 is the mean of a relevant reference population and 10 is the standard deviation (SD) of that population. For example a score of 40 is one SD lower than the mean of the reference population where as a score of 60 is one SD higher than the mean of the reference population. Thus a score of 60 is one standard deviation above the average referenced population. This could be a desirable or undesirable outcome, depending upon the concept being measured.
Change from Baseline Foot and Ankle Ability Measure at 12 weeks | Collected preoperatively and 12 weeks postoperatively
  Foot and Ankle Ability Measure (FAAM), a Patient Reported Outcome survey used widely in orthopaedic Foot and Ankle literature, will be obtained and reported in points. Scores range from 0% (least function) to 100% (most function).

SECONDARY OUTCOMES:
Pain Score | Assessed preoperatively and at 2 hours and 3, 6 and 12 weeks postoperatively
  Patients will score their pain on a Visual Analog pain scale (VAS) (0-10)
Malleolar circumference | Collected at 6 weeks and 12 weeks postoperatively
  bilateral malleolar circumference in cm will be measured by blinded physical therapists
Calf girth | Collected at 6 weeks and 12 weeks postoperatively
  bilateral calf girth in cm will be measured by blinded physical therapists
Mobility | Collected at 6 weeks and 12 weeks postoperatively
  Mobility, via timed up and go test in seconds, will be measured by blinded physical therapists. Patients will be seated in a chair and the time to rise, walk 10 feet, turn, walk back to the chair and sit down will be recorded in seconds.
Ankle range of motion | Collected at 6 weeks and 12 weeks postoperatively
  ankle range of motion (flexion, extension, inversion, eversion) will be measured in degrees with goniometer by blinded physical therapists
Fatigability | Collected at 6 weeks and 12 weeks postoperatively
  Utilizing a biodex machine, fatigability or total work in foot pounds, will be measured by blinded physical therapists
Proximal and distal lower extremity strength | Collected at 6 weeks and 12 weeks postoperatively
  proximal and distal lower extremity strength, via handheld dynamometer, in lb will be measured by blinded physical therapists
Single-limb stance time | Collected at 6 weeks and 12 weeks postoperatively
  Single-limb stance time (seconds) will be measured by blinded physical therapists
Y-balance test scores | Collected at 6 weeks and 12 weeks postoperatively
  Y-balance test composite score (%) will be measured by blinded physical therapists. For this test, the length of the extremity is measured and the patient reaches the extremity for the longest distance in three planes (anterior, posteriomedial, posterolateral) and the greatest distances achieved are recorded. The score is obtained by the sum of the greatest distances reached in each plane divided by 3x the limb length.
Limb pH | Recording will start immediately after placement of the probe and will continue intraoperatively and for 2 hours postoperatively
  a VersaFlex® pH catheter from the Covidien pH monitoring kit will be placed in the anterior compartment of the operative leg via small incision and the Digitrapper® Recorder will measure and record continuous intramuscular pH

CONTACTS AND LOCATIONS:
Overall Officials: Lara Atwater, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Omeroglu H, Gunel U, Bicimoglu A, Tabak AY, Ucaner A, Guney O. The relationship between the use of tourniquet and the intensity of postoperative pain in surgically treated malleolar fractures. Foot Ankle Int. 1997 Dec;18(12):798-802. doi: 10.1177/107110079701801208. PMID 9429882
- [Background] Konrad G, Markmiller M, Lenich A, Mayr E, Ruter A. Tourniquets may increase postoperative swelling and pain after internal fixation of ankle fractures. Clin Orthop Relat Res. 2005 Apr;(433):189-94. doi: 10.1097/01.blo.0000151849.37260.0a. PMID 15805957
- [Background] Younger AS, Kalla TP, McEwen JA, Inkpen K. Survey of tourniquet use in orthopaedic foot and ankle surgery. Foot Ankle Int. 2005 Mar;26(3):208-17. doi: 10.1177/107110070502600305. PMID 15766423
- [Background] Hung M, Baumhauer JF, Licari FW, Voss MW, Bounsanga J, Saltzman CL. PROMIS and FAAM Minimal Clinically Important Differences in Foot and Ankle Orthopedics. Foot Ankle Int. 2019 Jan;40(1):65-73. doi: 10.1177/1071100718800304. Epub 2018 Oct 4. PMID 30282469
- [Background] Wilgis EF. Observations on the effects of tourniquet ischemia. J Bone Joint Surg Am. 1971 Oct;53(7):1343-6. No abstract available. PMID 5114697
- [Background] Cushing H. Pneumatic tourniquets: with especial reference to their use in craniotomies: Medical news; 1904.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT05445960/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT05445960/ICF_001.pdf